CLINICAL TRIAL: NCT04986826
Title: Exercise Effect on Transthyretin Stability in Master Athletes and Patients With Transthyretin Amyloidosis
Brief Title: Exercise Effect on Transthyretin Stability
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Ahmad Masri, Principal Investigator, Oregon Health and Science University
Other Study IDs: 00023050
Record Dates: First submitted 2021-07-21; First posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Amyloidosis Transthyretin; Athlete Heart
Keywords: exercise; amyloidosis
MeSH Terms: conditions — Amyloid Neuropathies, Familial; Motor Activity; Amyloidosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy master athletes
- Genotype positive phenotype negative transthyretin amyloidosis
- Phenotype positive transthyretin amyloidosis

SUMMARY:
The goal of this study to investigate if exercise predisposes to transthyretin instability. The investigators will evaluate the effect of exercise on transthyretin biochemistry.

DETAILED DESCRIPTION:
This is an investigator initiated observational study, designed to study the effect of exercise on transthyretin stability in three main populations: Group 1: healthy master athletes who are 60 years or older. Group 2: Genotype positive (G+) cardiac phenotype negative (P-) patients with variant ATTR (i.e. carriers without evidence of disease). Group 3: Patients with ATTR CA who have not been on a stabilizer (tafamidis) within the last 14 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

General inclusion criteria: patients should be able to exercise on a treadmill or a bike, willing to consent to the study procedures and willing to return to site during the follow up period of 72 hours for repeated blood and urine collection

Specific inclusion criteria:

* Group 1: Subjects must be at least 60 years of age and meet the master athlete definition of: athletes engaged in cycling ≥8 hours per week or running ≥6 hours per week or triathlon training (combination of swimming, cycling, running) ≥8 hours per week, or equivalent sports activities, for at least 6 months prior to enrollment.
* Group 2: Genotype positive (G+) cardiac phenotype negative (P-) patients with variant ATTR (i.e. carriers without evidence of disease)
* Group 3: Patients with ATTR CA who have not been on a stabilizer (tafamidis) within the last 14 days prior to enrollment.

Exclusion Criteria:

Taking diflunisal or daily non-steroidal anti-inflammatory drugs (NSAIDs) use within 2 weeks.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Master athletes without evidence of transthyretin amyloidosis. Genotype positive phenotype negative transthyretin amyloidosis, and phenotype positive transthyretin amyloidosis.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-11-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in percent transthyretin stability assay | Change from baseline to 72 hours post-exercise
  Transthyretin stability will be measured and expressed as a percentage

SECONDARY OUTCOMES:
Plasma transthyretin level | Change from baseline to 72 hours post-exercise
  Plasma transthyretin level will be measured
Plasma transthyretin fragments | Change from baseline to 72 hours post-exercise
  Plasma transthyretin fragments will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No